CLINICAL TRIAL: NCT01975558
Title: The Radiation Metabolic Signature of Patient Undergoing Radiotherapy. A Pilot Study
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 181/11
Record Dates: First submitted 2013-09-04; First posted 2013-11-04 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, sebum, saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group A: Control group. The group will undergo blood, urine, sebum, and saliva sampling.
  Interventions: Biological: Sampling at baseline, one week after baseline, two weeks after baseline
- Breast cancer B: Breast cancer (60 Gy). The group will undergo blood, urine, sebum, and saliva sampling within the irradiation field.
  Interventions: Biological: Sampling at baseline, during radiotherapy and after
- Breast cancer C: Breast cancer (60 Gy). The group will undergo blood, urine, sebum, and saliva sampling outside of the irradiation field, e.g. at the arm.
  Interventions: Biological: Sampling at baseline, during radiotherapy and after

INTERVENTIONS:
Biological: Sampling at baseline, one week after baseline, two weeks after baseline
  Groups: Control group A
Biological: Sampling at baseline, during radiotherapy and after
  Groups: Breast cancer B; Breast cancer C

SUMMARY:
Rationale: Local radiotherapy applied in the treatment of tumors changes the metabolic profile in the exposed area and/or systemically and specific radiation biomarkers can be identified in the respective matrices.

Purpose: This is a pilot study to verify in humans the results obtained from two animal models exposed to ionizing gamma-radiation. The classification of patients results from the treatment volume of radiotherapy for cancer disease. Two patient groups with breast cancer undergoing high-dose radiotherapy are selected and compared to control group of age matched healthy women.

DETAILED DESCRIPTION:
Background

Humans are exposed to ionizing radiation from several sources. Gamma-radiation exposure induces thereby both short- and long-term adverse effects. The radiation injuries to be expected in humans in the acute stage (days to some weeks after radiation exposure) correlate with the radiation dose that the individual has received. With very high doses gastrointestinal syndrome leads to death within a few days. The survival of the individual in the acute stage is therefore dramatically dependent on the rapid application of suitable therapies. It is decisive here to identify in the shortest possible time those persons who have been exposed to a critical radiation dose and to estimate the dose received in order to apply an adequate therapy. There are no satisfying test methods available today, which would enable the mass screening for radiation injury.

Furthermore to identify changes in the local or systemic human metabolic fingerprint, which are useful for the prediction of the individual sensitivity of patients to radiotherapy and / or lead to a better understanding of the molecular mechanisms involved in radiotherapy.

Objective

Primary: The primary endpoint is to affirm the results from the animal model in radiation metabolomics in human radiotherapy treatment.

Secondary: The secondary endpoints are to find new potential biomarkers for radiation biodosimetry in humans and to identify changes in the different sequences in measuring from local (sebum) and systemic (blood, saliva and urine) material.

Methods

Gas chromatographic separation and mass spectrometric detection of the metabolites present in a given matrix (urine, saliva, plasma, sebum).

ELIGIBILITY:
Radiotherapy: cancer treatment with total doses of more than 30 Gy, single fraction dose of at least 1.8 Gy/die. Big treatment/target volume. Age over 50 years, according to postmenopausal status. No simultaneous chemotherapy in breast cancer patients. For the control group: healthy volunteers (women), age over 50 years, according to postmenopausal status; no previous chemo - and cancer therapy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty patients with breast cancer. Ten healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in radiation metabolites | During radiation treatment, expected to be ca. 5 weeks
  To affirm the results from animal model in radiation metabolomics in human radiotherapy treatment.

SECONDARY OUTCOMES:
New potential biomarkers for radiation biodosimetry | During and after radiation treatment (at baseline, week 1,5 + 6, 8 weeks after therapy end)
  To find new potential biomarkers for radiation biodosimetry in humans and to identify changes in different sequences in measuring from local and systemic material.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Loessl, MD, Study Chair — Dept. of Radiation Oncology, University Hospital, Inselspital Bern
Locations (1):
- Department of Radio-Oncology, Bern University Hospital, Bern, Switzerland